CLINICAL TRIAL: NCT03316274
Title: Phase 1 Study to Evaluate the Safety, Feasibility and Immunologic Correlatives of Intra-lesional Nivolumab Therapy for Limited Cutaneous Kaposi Sarcoma
Brief Title: Intra-lesional Nivolumab Therapy for Limited Cutaneous Kaposi Sarcoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17872; NCI-2018-02529 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); P30CA082103 (NIH)
Record Dates: First submitted 2017-09-29; First posted 2017-10-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Kaposi Sarcoma; HIV/AIDS; Immunosuppression
MeSH Terms: conditions — Sarcoma, Kaposi; Acquired Immunodeficiency Syndrome | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nivolumab (Cohort A-Safety) (Experimental): Participants will receive a 10mg (or 1 mL) injection into a single KS lesion in the skin, every 2 weeks for 4 doses.
  Interventions: Drug: Nivolumab
- Nivolumab (Cohort B-Expansion) (Experimental): Participants from Cohort A with at least 1 lesion that is left untreated and additional participants receive injections in into up to 2 KS lesions in the skin, every 2 weeks for 4 doses. The injected volume will not exceed 10 mg (or 1 mL) each time. Lesions will be evaluated at week 26, and participants with lesion improvement may enroll in Cohort B-PLUS to receive additional injections.
  Interventions: Drug: Nivolumab
- Nivolumab (Cohort B-PLUS) (Experimental): Participants in Cohort B whose injected lesions achieved partial response or complete response by week 26 and who did not experience any serious adverse events, are permitted to receive additional injections up to 4 residual KS lesions (total volume 10 mg in 1 mL) every 2 weeks for up to 4 additional doses. Lesions will be assessed again after 26 weeks.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Given via intralesional injection
  Other Names: Nivolumab Injection; Opdivo

SUMMARY:
Infection with Kaposi sarcoma herpesvirus (KSHV, or human herpesvirus-8 (HHV-8)) causes Kaposi sarcoma (KS). These virally associated diseases occur more frequently in HIV-infected individuals, but can also be found in HIV-uninfected population. Evolution of immunosuppressive mechanisms presumably plays a permissive role in the development, progression and recurrence of these virus-associated cancers and pre-cancers. Currently, available treatment options for these lesions are imperfect and there is no clear treatment for patients with limited cutaneous Kaposi sarcoma (KS). Radiation and injection of vinblastine both have side effects that may not be acceptable. Nivolumab has been used to treat more extensive KS when given intravenously. To the best of the investigator's knowledge, this is the first study to evaluate the safety of intra-lesional injections of nivolumab in patients with KS.

DETAILED DESCRIPTION:
This is a single-center, phase I safety/expansion trial of nivolumab in HIV-infected (with stable, treated HIV on cART) and HIV-uninfected patients with limited cutaneous KS.

PRIMARY OBJECTIVES:

- To determine the safety and tolerability of four intra-lesional injections of nivolumab given every two weeks to treat KS. They will be assessed by NCI Common Terminology Criteria for Adverse Events version 5 (NCI CTCAE v. 5).

SECONDARY OBJECTIVES:

* To determine the changes in cytotoxic T cells and regulatory T cells in the lesions as determined by immunohistochemistry and flow cytometry.
* To determine the changes in cytotoxic T cells and regulatory T cells in the peripheral blood as determined by flow cytometry.
* To determine the changes in PD-1/PD-L1 expression as determined by immunohistochemistry in lesions.

OUTLINE:

Participants with treatment-experienced KS will be enrolled into Cohort A (initial safety cohort). If there are no grade 3 or higher adverse events, enrollment into the expansion cohort (Cohort) B will be available to participants with either treatment-experienced or treatment-naïve KS, including those previously enrolled in the safety cohort.

Patients will receive one intra-lesional injection of nivolumab into one cutaneous KS lesion every 2 weeks for up to a total of 4 doses until completed or intolerable toxicity, request to withdraw, or withdrawal per the Principal Investigator. Participants will be followed for an additional 5 months after completing the 4 treatment doses.

ELIGIBILITY:
Inclusion Criteria:

1. For screening: Participants must have histologically confirmed KS with active cutaneous disease and have less than 25 lesions. For enrollment: Participants must have histologically confirmed KS in the research skin biopsy performed during the screening visit.
2. Participants must have measurable cutaneous KS disease, defined as 1 or more marker lesion that is bi-dimensionally measurable, and >=0.5cm in shortest dimension. These measurable lesions must not have received previous local radiation, surgical, or intralesional cytotoxic therapy that would prevent response assessment. Note: Participants may eligible even if some KS lesions that have previously been treated with local therapy, as long as other untreated KS lesions are measurable as defined in the protocol.
3. For the initial safety cohort (cohort A), participants have to be treatment-experienced, i.e. at least one of the KS skin lesions has been persisted despite having been treated with:

   * systemic chemotherapy; OR
   * 1 or more topical therapy, local radiation, surgery, or intra-lesional cytotoxic therapy.

   For the expansion cohort (cohort B), participants can be either treatment-experienced or treatment-naïve.

   For the extension cohort (cohort B-plus), participants are from the expansion cohort above (cohort B) who have achieved partial response (PR) or complete response (CR) in their injected KS lesion at week 26 or later.
4. Age >= 18 years.
5. If human immunodeficiency virus (HIV)-infected, participants must have:

   * HIV-1 infection, documented by any federally approved, licensed HIV rapid test performed in conjunction with screening (or ELISA, test kit, and confirmed by Western blot or other approved test). Alternatively, this documentation may include a record demonstrating that another physician has documented the participant's HIV status based on either: 1) approved diagnostic tests, or 2) the referring physician's written record that HIV infection was documented, with supporting information on the participant's relevant medical history and/or current management of HIV infection
   * CD4 >= 350 cells/mm3
   * HIV-1 viral load below the limit of detection by commercial assays (<75 copies/mL).
   * Participants MUST receive appropriate care and treatment for HIV infection, including antiretroviral medications when clinically indicated, and should be under the care of a physician experienced in HIV management. Participants should be documented to be on an effective combination anti-retroviral (ART) regimen, generally a 3-drug regimen based on Department of Health and Human Services (DHHS) treatment guidelines by a licensed health care provider. Participants will be eligible regardless of antiretroviral medication (including no antiretroviral medication) provided there is no intention to initiate therapy or the regimen has been stable for at least 4 weeks with no intention to change the regimen within 12 weeks following enrollment.
6. If HIV-uninfected, participants must have documentation of a negative HIV result by any federally approved, licensed HIV test within the last 12 months.
7. Adequate organ function defined as follows:

   1. Leukocytes > 3,000/microliter (mcL).
   2. Absolute neutrophil count > 1,000/mcL.
   3. Hemoglobin > 10 g/dL.
   4. Platelets > 100,000/mcL.
   5. Total bilirubin within normal institutional limits.
   6. Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) < 2.5 X institutional upper limit of normal (ULN)
   7. Alanine aminotransferase (ALT)/ serum glutamic-pyruvic transaminase (SGPT) < 2.5 X institutional ULN
   8. Creatinine < 1.5 X institutional ULN
8. Participants must be purified protein derivative (PPD) negative. Alternatively, the QuantiFERON-TB Gold In-Tube (QFT-GIT) assay (Cellestis Limited, Carnegie, Australia) can be used. An individual is considered positive for M. tuberculosis (TB) infection if the Interferon (IFN)-gamma response to TB antigens is above the test cut-off (after subtracting the background IFN-gamma response in the negative control). The result must be obtained within 12 months prior to enrollment. PPD positive (or QuantiFERON assay positive) participants are permitted if prophylaxis has been completed prior to enrollment.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of <=1 (Karnofsky >= 70%).
10. The effects of nivolumab on the developing fetus are unknown. Therefore, only the following patients should be enrolled:

    1. Woman of child-bearing potential (WOCBP), defined as a sexually mature woman who has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries)) or, has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time during the preceding 24 consecutive months} must have negative serum pregnancy test within 7 days before starting study treatment in WOCBP and willingness to adhere to acceptable forms or birth control (a physician-approved contraceptive method (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner).

       WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 6 months after the last dose.

       Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study (including the time after last dose previously mentioned), she (or the participating partner) should inform the treating physician immediately.
    2. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product.

Exclusion Criteria:

1. Prior systemic KS-directed treatments or investigational modalities <= 5 half-lives or 4 weeks, whichever is shorter, prior to starting study drug or who have not recovered from side effects of such therapy to grade 1 or less.
2. Presence of any visceral KS (including KS-associated lymphedema) requiring systemic chemotherapy. This includes, but not limited to, any symptomatic visceral KS or asymptomatic pulmonary KS.
3. Hypersensitivity to nivolumab or any of its excipients.
4. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
5. Opportunistic infection within the last 3 months.
6. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
7. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent. This does not apply to participants in the extension cohort (cohort B-plus).
8. Active systemic immunosuppressive therapy.
9. The use of prednisone or equivalent 10mg or greater a day that cannot be discontinued with more than 7 consecutive days of steroids within the prior 2 weeks.
10. Prior organ allograft or allogeneic transplantation, if the transplanted tissue is still in place.
11. Unstable angina, significant cardiac arrhythmia, or New York Heart Association (NYHA) class 3 or 4 congestive heart failure.
12. Major surgery ≤ 2 weeks prior to starting a study drug or who have not recovered from side effects of such therapy.
13. Any significant medical condition, laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
14. Any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number participants with Dose Limiting Toxicities (DLT) (Cohort A) | 6 months
  The number of participants with DLTs will defined as treatment-related, grade 3-5 adverse events assessed using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Maximum Tolerated Dose (MTD) (Cohort A) | 6 months
  The MTD is defined as the dose at which no more than 1/6 patients experience a DLT

SECONDARY OUTCOMES:
Median percent change in absolute CD3 cells (CD3+) / CD4+ cells | 6 months
  Treatment induced, tumor infiltrating immune cells will be evaluated in pre-treatment and post-treatment tissue via immunohistochemistry (IHC).
Median percent change in cytotoxic T cells with CD8 surface protein (CD8+) T cells /Granzyme+ T cytotoxic T cells | 6 months
  Treatment induced, tumor infiltrating immune cells will be evaluated in pre-treatment and post-treatment tissue via immunohistochemistry (IHC).
Median percent change in CD56+ natural killer (NK) cells | 6 months
  Treatment induced, tumor infiltrating immune cells will be evaluated in pre-treatment and post-treatment tissue via immunohistochemistry (IHC).
Median percent change in CD4+FOXP3-effector T cells | 6 months
  Treatment induced, tumor infiltrating immune cells will be evaluated in pre-treatment and post-treatment tissue via immunohistochemistry (IHC).
Median percent change in CD4+FOXP3+regulatory T cells | 6 months
  Treatment induced, tumor infiltrating immune cells will be evaluated in pre-treatment and post-treatment tissue via immunohistochemistry (IHC).
Changes in Circulating plasma cytokines | 6 months
  Circulating plasma cytokines will be evaluated in pre-treatment and post-treatment
Changes in frequency of circulating activated T cells in the peripheral blood | 6 months
  Frequency of circulating activated T cells in the peripheral blood induced by intra-lesional nivolumab therapy will be assessed via flow cytometry
Median change in number of circulating activated T cells in the peripheral blood | 6 months
  Changes in number of circulating activated T cells in the peripheral blood induced by intra-lesional nivolumab therapy will be assessed via flow cytometry
Changes in PD-1 expression as determined by immunohistochemistry in lesions | 6 months
  Changes in PD-L1 expression induced by intra-lesional nivolumab therapy will be assessed via IHC, using commercially available PD-1 antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-ching Wang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT03316274/ICF_000.pdf